CLINICAL TRIAL: NCT05592158
Title: Evaluation of the Effectiveness of an Amnion-chorion Membrane for Alveolar Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Muhammad Saleh, Clinical Assistant Professor, Periodontics and Oral Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00208140
Record Dates: First submitted 2022-10-07; First posted 2022-10-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Healing Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (Experimental): Amnion-chorion membrane with collagen plug
  Interventions: Procedure: Socket preservation
- Control (Active Comparator): Collagen plug
  Interventions: Procedure: Socket preservation

INTERVENTIONS:
Procedure: Socket preservation — After tooth extraction, the socket will be filled with a collagen plug and covered with an amnion-chorion membrane.

SUMMARY:
This study will examine whether adding an amnion-chorion membrane on top of the traditionally used collagen plug will lead to more bone formation compared to the collagen plug only.

DETAILED DESCRIPTION:
Bone grafts and membranes are commonly placed to increase the amount of bone right after tooth extraction and before placing a dental implant. The primary objective of this study is to study the effect of a human amnion-chorion membrane (ACM) in an exposed-barrier ridge preservation technique to a control group without utilizing a ACM.

30 patients requiring a front tooth extraction will be recruited and randomized to receive bone grafting with or without an ACM.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 20 to 80 years.
2. Patients must require tooth extraction (for incisors, canines and premolars) as a result of caries, periodontal disease, tooth fracture or deemed unrestorable.
3. Socket should be free of infection, less than 5mm of dehiscence
4. Patients interested in implant placement following tooth extraction.

Exclusion Criteria:

1. Allergies or hypersensitivities to study related medications such as chlorhexidine.
2. Hematologic disorders/blood dyscrasias.
3. Active infectious diseases of any kind.
4. Liver or kidney dysfunction/failure.
5. Uncontrolled diabetes (HbA1c > 8).
6. Active cancer treatment - such as active chemotherapy or radiation therapy.
7. Taking medications that will affect their bone healing (for example, bisphosphonates).
8. Metabolic bone diseases that affect bone healing such as osteoporosis.
9. Pregnant or lactating women (self-reported).
10. Smoke 10 or more cigarettes per day (self-reported).
11. Poor oral hygiene.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Clinical alveolar ridge dimension changes | 4 months
  Clinically measured alveolar ridge dimension changes in mm using calibers
Digital alveolar ridge dimension changes | 4 months
  Digitally measured alveolar ridge dimension changes in mm2 using CBCT

SECONDARY OUTCOMES:
Histological bone density. | 4 months
  Histomorphometry.
Presence of bone turnover proteins. | 4 months
  Immunohistochemistry.
Implant survival-Clinical | 6 months
  Clinically assessed by torque test using a torque wrench, measured in N/cm.
Implant survival-Radiographic | 6 months
  Radiographically assessed through any signs of radiolucency around the implant.
Esthetic restorative outcomes. | 6 months
  Clinical changes in hard tissue based on the PES score

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Saleh, BDS, MSD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No